CLINICAL TRIAL: NCT05271409
Title: A Phase III, Randomized, Double-blind, Placebo-controlled, Multicenter Study to Evaluate the Efficacy, Safety, Pharmacokinetics, and Pharmacodynamics of Satralizumab as Monotherapy or in Addition to Baseline Therapy in Patients With Myelin Oligodendrocyte Glycoprotein Antibody-associated Disease (MOGAD)
Brief Title: A Study to Evaluate the Efficacy, Safety, Pharmacokinetics, and Pharmacodynamics of Satralizumab in Participants With Myelin Oligodendrocyte Glycoprotein Antibody-associated Disease
Acronym: Meteoroid
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WN43194; 2021-003192-34 (EudraCT Number); 2023-507196-22-00 (EU CTIS Number)
Record Dates: First submitted 2022-02-28; First posted 2022-03-09 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Myelin Oligodendrocyte Glycoprotein Antibody-Associated Disease (MOGAD)
MeSH Terms: conditions — Myelin Oligodendrocyte Glycoprotein Antibody-Associated Disease | interventions — satralizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Satralizumab (Experimental): In the DB treatment period, participants will receive satralizumab at Weeks 0, 2, 4 (loading doses) and maintenance doses every 4 weeks (Q4W) thereafter. In the OLE period, all participants will receive open-label treatment with satralizumab. Additional adolescent participants will be directly enrolled in the OLE period to receive satralizumab.
  Interventions: Drug: Satralizumab
- Placebo (Placebo Comparator): In the DB treatment period, participants will receive satralizumab matching placebo at Weeks 0, 2, 4 (loading doses) and maintenance doses Q4W thereafter. In the OLE period, all participants will receive open label treatment with satralizumab.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Satralizumab — Study drug will be administered by subcutaneous (SC) injection in the abdominal or femoral region after all other study-related procedures have been performed at a site visit.
  Arms: Satralizumab
Other: Placebo — Placebo will be administered by SC injection in the abdominal or femoral region after all other study-related procedures have been performed at a site visit.
  Arms: Placebo

SUMMARY:
The main objective of this study is to evaluate the efficacy of satralizumab compared with placebo based on time from randomization to the first occurrence of an adjudicated MOGAD relapse in the double-blind (DB) treatment period. Participants who experience an adjudicated relapse or complete the DB period can enter open-label extension (OLE) period. After the primary clinical cutoff date (CCOD), additional adolescent participants may be enrolled directly into the OLE period.

ELIGIBILITY:
Inclusion criteria

* Participants who are aged >=12 years at the time of signing Informed Consent Form
* Confirmed diagnosis of MOGAD with a history of >=1 MOGAD relapse in the 12 months prior to screening or >=2 attacks in the 24 months prior to screening
* Expanded Disability Status Scale (EDSS) score of 0-6.5 at screening
* High-contrast visual acuity (HCVA) better than 20/800 in each eye at screening
* Participants receiving either no or ongoing chronic immunosuppressant treatment (IST) for MOGAD at the time of screening
* For women of childbearing potential: participants who agree to remain abstinent or use adequate contraception during the treatment period and for at least 3 months after the final dose of satralizumab

Exclusion criteria

* Presence of aquaporin-4-antibodies immunoglobin G (AQP4-IgG) in the serum
* History of anti-N-methyl-d-aspartate receptor (NMDAR) encephalitis
* Any concomitant disease other than MOGAD that may require treatment with ISTs or oral corticosteroids (OCS) or intravenous (IV) corticosteroids at doses > 20 milligrams (mg) prednisone equivalent per day for >21 days during the study
* Participants who are pregnant or breastfeeding, or intending to become pregnant during the study or within 3 months after the final dose of satralizumab
* Participants with active or presence of recurrent bacterial, viral, fungal, mycobacterial infection, or other infection at baseline
* Participants with evidence of latent or active tuberculosis (excluding patients receiving chemoprophylaxis for latent tuberculosis infection)
* Participants with positive screening tests for hepatitis B and C
* Receipt of live or live attenuated vaccine within 6 weeks prior to baseline
* History of severe allergic reaction to a biologic agent

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2022-08-30 (Actual); Primary Completion 2025-11-20 (Actual); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Time From Randomization to the First Occurrence of a MOGAD Relapse in the DB Treatment Period, as Determined by an Adjudication Committee (CEC) | Up to approximately 44 months

SECONDARY OUTCOMES:
Annualized Rate of Adjudicated MOGAD Relapses | Up to approximately 44 months
Annualized Rate of Active Lesions on Magnetic Resonance Imaging (MRI) of the Neuroaxis | Up to approximately 44 months
Proportion of Participants Receiving Rescue Therapy | Up to approximately 44 months
Annualized Rate of Inpatient Hospitalizations | Up to approximately 44 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (82):
- United States (23):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic- Scottsdale, Scottsdale, Arizona
  - University of California Irvine - Manchester Pavilion, Irvine, California
  - University of Colorado - Anschutz Medical Campus (University of Colorado Health Sciences Center), Aurora, Colorado
  - Medstar Georgetown University Hospital, Washington D.C., District of Columbia
  - University of Florida College of Medicine Gainesville, Gainesville, Florida
  - Nemours Children's Clinic - of the Nemours Foundation, Jacksonville, Florida
  - Meridian Clinical Research, LLC, Savannah, Georgia
  - Northwestern University, Chicago, Illinois
  - Consultants in Neurology Ltd, Northbrook, Illinois
  - Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Memorial Healthcare Institute for Neurosciences and Multiple Sclerosis, Owosso, Michigan
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - NYU Langone, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - OhioHealth Research Institute, Columbus, Ohio
  - Premier Neurology, Greenville, South Carolina
  - Baylor College of Medicine, Houston, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (9):
  - Brain and Mind Research Institute, Camperdown, New South Wales
  - John Hunter Hospital, New Lambton, New South Wales
  - Sydney Children's Hospital, Randwick, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Box Hill Hospital, Box Hill, Victoria
  - Monash Medical Centre, Clayton, Victoria
  - St Vincent's Hospital Melbourne, Fitzroy, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Perron Institute for Neurological and Translational Science, Nedlands, Western Australia
- Brazil (4):
  - Instituto de Neurologia de Curitiba, Curitiba, Paraná
  - Instituto do Cerebro do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul
  - Centro de Pesquisas Clinicas, São Paulo, São Paulo
  - Hospital Universitario Gaffree e Guinle, Rio de Janeiro
- Canada (5):
  - London Health Sciences Centre Uni Campus, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Unity Health Toronto - St. Michael's Hospital, Toronto, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - MUCH - Montreal Neurological Institute & Hospital, Montreal, Quebec
- France (3):
  - Hopital Pierre Wertheimer, Bron
  - CH de Bicêtre, Le Kremlin-Bicêtre
  - CHU de Toulouse - Hôpital Purpan, Toulouse
- Germany (7):
  - NeuroCure Clinical Research Center (NCRC), Berlin
  - St. Josef-Hospital, Klinik für Neurologie, Bochum
  - Vestische Kinder- und Jugendklinik Datteln, Datteln
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Neurology UKSH Campus Kiel, Kiel
  - Universitätsklinikum Mannheim, Mannheim
  - Klinikum Großhadern, LMU, Munich
- Hadassah University Hospital Ein Kerem, Jerusalem, Israel
- Italy (7):
  - Ospedale Pediatrico Bambino Gesù, Rome, Lazio
  - IRCCS Ospedale San Raffaele, Milan, Lombardy
  - Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan, Lombardy
  - Fondazione Istituto Neurologico Mondino IRCCS, Pavia, Lombardy
  - Azienda Sanitaria Ospedaliera S. Luigi Gonzaga, Orbassano, Piedmont
  - AOU Policlinico V. Emanuele - P.O G. Rodolico, Catania, Sicily
  - Azienda Ospedaliera Universitaria Integrata Verona, Verona, Veneto
- Japan (14):
  - Chiba University Hospital, Chiba
  - Kyushu University Hospital, Fukuoka
  - Southern Tohoku Medical Clinic, Fukushima
  - Kobe University Hospital, Hyōgo
  - Kitasato University Hospital, Kanagawa
  - Tohoku University Hospital, Miyagi
  - Tohoku Medical and Pharmaceutical University Hospital, Miyagi
  - The University of Osaka Hospital, Osaka
  - Saitama Medical Center, Saitama
  - The Jikei University Hospital, Tokyo
  - Juntendo University Hospital, Tokyo
  - Tokyo Medical University Hospital, Tokyo
  - Keio University Hospital, Tokyo
  - Tokyo Women's Medical University Hospital, Tokyo
- Poland (6):
  - Wielospecjalistyczna Poradnia Lekarska Synapsis, Katowice
  - Szpital Uniwersytecki w Krakowie, Krakow
  - Centrum Medyczne "MEDYK", Rzeszów
  - Klinika Neurologii I Wydzialu Lekarskiego WUM w Warszawie, Warsaw
  - Instytut Pomnik Centrum Zdrowia Dziecka, Warsaw
  - SPSK nr 1, Zabrze
- South Korea (3):
  - National Cancer Center, Goyang-si
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing